CLINICAL TRIAL: NCT01287364
Title: Psychometric Evaluation of a Novel Questionnaire Designed to Assess Patient Satisfaction With and Preference of Intranasal Corticosteroids Administered Via HFA Aerosol or Aqueous Suspension Used for the Treatment of Allergic Rhinitis
Brief Title: Evaluation of a Novel Questionnaire to Assess Patient Satisfaction With and Preference of Intranasal Corticosteroids for the Treatment of Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 060-301
Record Dates: First submitted 2011-01-26; First posted 2011-02-01 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Perennial Allergic Rhinitis
Keywords: perennial allergic rhinitis; PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Nasal Sprays; Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ciclesonide HFA followed by mometasone (Experimental): ciclesonide hydrofluoroalkane (HFA) nasal aerosol 80 μg once daily in first intervention period, followed by a 7-14 day washout period, after which the second intervention of mometasone nasal inhalation 200 μg once daily will be administered.
  Interventions: Drug: ciclesonide hydrofluoroalkane (HFA) nasal aerosol; Drug: mometasone nasal inhalation
- mometasone followed by ciclesonide HFA (Active Comparator): mometasone nasal inhalation 200 μg once daily in first intervention period followed by a 7-14 day washout period after which the second intervention of ciclesonide hydrofluoroalkane (HFA) nasal aerosol 80 μg once daily will be administered
  Interventions: Drug: ciclesonide hydrofluoroalkane (HFA) nasal aerosol; Drug: mometasone nasal inhalation

INTERVENTIONS:
Drug: ciclesonide hydrofluoroalkane (HFA) nasal aerosol — ciclesonide hydrofluoroalkane (HFA) nasal aerosol 80 μg once daily for one week.
Drug: mometasone nasal inhalation — mometasone nasal inhalation 200 μg once daily for one week
  Other Names: Nasonex®

SUMMARY:
This is an open-label, randomized, multicenter, 2-way crossover study in subjects 12 years or older with perennial allergic rhinitis (PAR) to evaluate the psychometric properties of a novel-patient administered assessment of treatment satisfaction with and preference of an Internasal Corticosteroid (INCS)

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, 2-way crossover study in subjects 12 years or older with perennial allergic rhinitis (PAR) to evaluate the psychometric properties of a novel-patient administered assessment of treatment satisfaction with and preference of an INCS. Subjects will be randomized to 1 of 2 treatment sequences:

Sequence 1: Treatment Period 1 = ciclesonide hydrofluoroalkane (HFA) nasal aerosol 80 μg once daily; Treatment Period 2 = mometasone nasal inhalation 200 μg once daily

Sequence 2: Treatment Period 1 = mometasone nasal inhalation 200 μg once daily; Treatment Period 2 = ciclesonide HFA nasal aerosol 80 μg once daily

Total study participation will be approximately 8 weeks including a 3-week screening/baseline phase, a 1-week treatment period, a 1- to 2- week washout phase between treatments, a second 1-week treatment period consisting of the alternate treatment, and an additional 1-week follow up period after the last dose of study drug to assess safety. Subjects are required to continue to meet eligibility criteria for the second treatment period.

Nasal symptoms will be evaluated daily from 7 days prior to the first dose of study drug in Treatment Period 1 through the last dose of study drug in Treatment Period 2. The Allergic Rhinitis Satisfaction and Preference (ARTSP) and other Modules from the Phase V® e-Health Outcomes Information System (Phase V Technologies, Wellesley MA) will be completed two times during each treatment period (before the first dose and on the day after the last dose) via the internet at the clinical site. Patient preference will be evaluated at the day after last dose only.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent and assent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Male or female 12 years and older at screening
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on screening physical examination, clinical laboratory results, and medical history.
* A history of PAR to a relevant perennial allergen (house dust mites, cockroach, molds, animal dander) for a minimum of two years immediately preceding screening. The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past, and require treatment with an INCS throughout the entire study period.
* At least one treatment for PAR during the 6 months prior to expected randomization was a nasal spray.
* A demonstrated sensitivity to at least one allergen known to induce PAR (house dust mites, animal dander, cockroach, and molds) based on a documented result with a standard skin-prick test either within 90 days prior to or at screening. A positive test is defined as a wheal diameter at least 3 mm larger than the negative control wheal for the skin-prick test. The subject's positive test for the allergen must be consistent with the medical history of PAR and the allergen must be present in the subject's environment throughout the study.
* Based upon subject's medical history, in the investigator's judgment, the subject is unlikely to have a seasonal allergy exacerbation during the study.
* Subject, if female ≤ 65 years of age, must have a negative serum pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: a. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for 30 days following completion of study participation. b.Barrier method of contraception, e.g., condom and/or diaphragm with spermicide while participating in the study. c.Abstinence.
* The subject must possess a degree of understanding of written English, in the opinion of the investigator that enables them to complete the Phase V® Technologies Inc. (PVT) Modules.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; or nasal ulcers or perforations. Surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the last 60 days prior to screening.
* Presently has nasal jewelry, has had a nasal piercing, or a history of nasal surgery (e.g., rhinoplasty, septoplasty) or trauma to the nasal cavity.
* Subject is, in the investigator's judgment, having a seasonal exacerbation at screening.
* Participation in any investigational drug trial within the 30 days preceding screening or planned participation in another investigational drug trial at any time during this study.
* A known hypersensitivity to any corticosteroid or any of the components in the formulations of ciclesonide or Nasonex.
* History of a respiratory infection or disorder (including, but not limited to, bronchitis, pneumonia, influenza, severe acute respiratory syndrome [SARS]) within the 14 days preceding screening.
* History of alcohol or drug abuse within 2 years preceding screening.
* History of a positive test for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta agonists and any controller drugs (e.g., theophylline, leukotriene antagonists, etc.); intermittent use (less than or equal to three uses per week) of inhaled short-acting beta-agonists is acceptable. Use of short-acting beta-agonists for exercise-induced bronchospasm is allowed.
* Expected use of any disallowed medications during the study period.
* Expected initiation of immunotherapy during the study period or planned dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to screening and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Non-vaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding screening.
* Expected initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Study participation by clinical site employees and/or their immediate relatives who reside in the same household.
* Study participation by more than one subject from the same household.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial: impaired hepatic function including alcohol related liver disease or cirrhosis; history of ocular disturbances, e.g., glaucoma or posterior subcapsular cataracts; any systemic infection; hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism) disease; gastrointestinal disease; malignancy (excluding basal cell carcinoma); current neuropsychological condition with or without drug therapy
* Any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with completion of the assessments as written.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Allergy and Asthma Associates of Southern California, Mission Viejo, California
  - Allergy & Asthma Medical Group & Research Center A.P.C., San Diego, California
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneappolis, Minnesota
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Sylvania Research Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciclesonide HFA Followed by Mometasone: ciclesonide hydrofluoroalkane nasal aerosol (HFA) 80 μg once daily in first intervention period, followed by a 7-14 day washout period, after which the second intervention of mometasone nasal inhalation 200 μg once daily will be administered.
Period: Overall Study
Arm/Group | Ciclesonide HFA Followed by Mometasone | Mometasone Followed by Ciclesonide HFA
Started | 94 | 91
Completed | 85 | 81
Not Completed | 9 | 10
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 5 | 5
Not completed — Other Reason | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide HFA Followed by Mometasone | Mometasone Followed by Ciclesonide HFA | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 12 | 21
  Between 18 and 65 years | 81 | 78 | 159
  >=65 years | 4 | 1 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (15.1) | 37.5 (14.6) | 38.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 56 | 121
  Male | 29 | 35 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 40
  Not Hispanic or Latino | 76 | 69 | 145
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 80 | 77 | 157
  Black or African American | 10 | 7 | 17
  Asian | 3 | 3 | 6
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 0 | 2 | 2
  Multiple | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction Subscales (Interference, Regimen Adaptation, Role Limitations, Sensory Impact, Regimen Difficulties, Burden, Hassle, Regimen Management, and Perceived Relief)Reliability Statistics
Description: Reliability for the nine treatment satisfaction subscales was established through internal consistency statistical analyses [Cronbach's alpha (raw and standardized) coefficients were calculated]. The correlation coefficients for these analyses ranged from 0.0 to 1.0, with higher coefficients indicating greater reliability. A coefficient of ≥ 0.7 was the standard for evidence of reliability.
Time Frame: Day 1 (Pre-treatment) through Day 7 Treatment Period 2
Population: Subjects from Treatment Sequence AB (ciclesonide nasal aerosol 74 mcg/mometasone nasal spray 200 mcg) and Treatment Sequence BA (mometasone nasal spray 200 mcg/ciclesonide nasal aerosol 74 mcg) were pooled. Validation was performed without regard to treatment, thus all observations were pooled.
Measure: Number; unit: ratio of variance
Groups:
- Average Cronbach's Alpha (Raw) Coefficients; Average Cronbach's Alpha (Standardized) Coefficients: Cronbach's alpha coefficient, which is a correlation coefficient ranging from 0.0 to 1.0 with higher coefficients indicating greater reliability. A coefficient of ≥ 0.7 was the standard for evidence of reliability.
Arm/Group | Average Cronbach's Alpha (Raw) Coefficients | Average Cronbach's Alpha (Standardized) Coefficients
Number analyzed (Participants) | 185 | 185
ratio of variance
  Interference | 0.971 | 0.972
  Regimen Adaptation | 0.932 | 0.932
  Role Limitations | 0.939 | 0.944
  Sensory Impact | 0.889 | 0.895
  Regimen Difficulties | 0.722 | 0.731
  Hassle | 0.918 | 0.928
  Burden | 0.937 | 0.938
  Regimen Management | 0.750 | 0.804
  Perceived Relief | 0.864 | 0.871

2. Primary Outcome: Discriminant Validity of Treatment Satisfaction Subscales Statistical Analyses Based on Baseline Reflective Total Nasal Symptom Score (rTNSS) Categories (Low, Medium, High)
Description: Discriminant validity tests whether the subscales differentiate among groups of respondents that differ on a pre-specified criterion, baseline rTNSS. Patients were assigned to baseline rTNSS categories of Low Symptoms(3.00 - 7.17; n = 62), Medium Symptoms (7.25 - 9.25; n = 61), or High Symptoms (9.33 - 12.00; n = 62). Reflective TNSS group served as the independent variable and the nine treatment satisfaction subscales were evaluated as dependent variables by analysis of variance models. Contrasts were tested between the Low and Medium Symptoms and the High and Low Symptom categories. Reflective TNSS group served as the independent variable and the nine treatment satisfaction subscales were evaluated as dependent variables by analysis of variance models. All of the treatment satisfaction subscales and satisfaction scales were scored from 0 (low satisfaction) to 100 (high satisfaction).
Time Frame: Day 1 (Pre-treatment) through Day 7 Treatment Period 1
Population: Baseline rTNSS was partitioned into tertile ranges and patients were assigned to Low (3.00 - 7.17; n = 62), Medium (7.25 - 9.25; n = 61), or High (9.33 - 12.00; n = 62) symptom groups.
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Low Symptoms: Patients were assigned to baseline rTNSS categories of Low Symptoms(3.00 - 7.17; n = 62). Results reported as difference in mean treatment satisfaction subscale score range 0-100 where higher represent greater satisfaction. TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval.
- Medium Symptoms: Patients were assigned to baseline rTNSS categories of Medium Symptoms (7.25 - 9.25; n = 61). Results reported as difference in mean treatment satisfaction subscale score range 0-100 where higher represent greater satisfaction. TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval.
- High Symptoms: Patients were assigned to baseline rTNSS categories of High Symptoms (9.33 - 12.00; n = 62). Results reported as difference in mean treatment satisfaction subscale score range 0-100 where higher represent greater satisfaction. TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval.
Arm/Group | Low Symptoms | Medium Symptoms | High Symptoms
Number analyzed (Participants) | 62 | 61 | 62
scores on a scale
  Interference | 78.726 (3.186) | 70.931 (3.160) | 59.018 (3.160)
  Regimen Adaptation | 60.764 (2.4575) | 59.491 (2.455) | 53.455 (2.455)
  Role Limitation | 87.141 (2.322) | 83.528 (2.303) | 73.269 (2.303)
  Regimen Difficulty | 85.940 (2.254) | 78.890 (2.235) | 71.676 (2.235)
  Sensory Impact | 67.934 (2.660) | 61.452 (2.638) | 53.742 (2.638)
  Hassle | 63.361 (3.725) | 49.839 (3.695) | 40.726 (3.695)
  Burden | 77.818 (2.606) | 76.109 (2.585) | 60.534 (2.585)
  Regimen Management | 80.949 (2.094) | 81.771 (2.077) | 72.192 (2.077)
  Perceived Relief | 56.066 (2.435) | 55.457 (2.415) | 50.054 (2.415)
  Overall Satisfaction | 73.189 (1.927) | 68.607 (1.911) | 59.407 (1.911)

3. Primary Outcome: Responsiveness Statistical Analysis of Treatment Satisfaction Subscales for Treatment Period 1 Versus Change in rTNSS From Baseline Categories (Low Change, Medium Change, or High Change)
Description: Analysis was conducted with one-sample t-tests on the treatment satisfaction subscale change scores for Treatment Period 1 against the test criterion of "no change" (ie, change score = 0)TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. TNSS values range from 0-12 (0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. All of the treatment satisfaction subscales and satisfaction scales were scored from 0 (low satisfaction) to 100 (high satisfaction).
Time Frame: Day 1 (pre-treatment) through Day 7 Treatment Period 1
Population: The rTNSS total period 1 change scores were partitioned into tertile ranges to form three groups: Low Change (-1.04 - -4.93; n = 60), Medium Change (-2.49 - -1.05; n = 62), and High Change (-7.57 - -2.50; n = 61).
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Low Change; Medium Change; High Change: rTNSS change scores were partitioned into three categories to form the independent variable - Low Change (0.70 to 1.85), Medium Change (2.08 to 1.74), or High Change (6.57 to 2.14) groups.
Arm/Group | Low Change | Medium Change | High Change
Number analyzed (Participants) | 60 | 62 | 61
scores on a scale
  Interference | 10.492 (2.458) | 15.836 (2.496) | 20.380 (2.922)
  Regimen Adaptation | 1.121 (2.531) | 12.121 (2.469) | 13.333 (3.199)
  Role Limitation | 9.764 (1.121) | 10.512 (1.721) | 12.440 (1.732)
  Regimen Difficulty | -1.083 (2.475) | 3.760 (2.579) | 2.083 (2.710)
  Sensory Impact | 12.667 (2.270) | 13.226 (2.702) | 19.475 (2.959)
  Hassle | 11.250 (3.114) | 17.742 (2.723) | 26.475 (3.660)
  Burden | 15.469 (2.223) | 16.331 (2.321) | 16.701 (2.809)
  Regimen Management | 8.042 (1.583) | 9.348 (1.820) | 9.027 (1.587)
  Perceived Relief | -2.917 (3.296) | 8.280 (2.840) | 12.705 (3.706)
  Overall Satisfaction | 7.201 (1.314) | 11.906 (1.479) | 14.735 (1.799)

4. Primary Outcome: Responsiveness Statistical Analysis of Treatment Satisfaction Subscales for Treatment Period 2 Versus Change in rTNSS From Baseline Categories (Low Change, Medium Change, or High Change)
Description: Analysis was conducted with one-sample t-tests on the treatment satisfaction subscale change scores for Treatment Period 2 against the test criterion of "no change" (ie, change score = 0)TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. TNSS values range from 0-12 (0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. All of the treatment satisfaction subscales and satisfaction scales were scored from 0 (low satisfaction) to 100 (high satisfaction).
Time Frame: Day 1 (pre-treatment) through Day 7 Treatment Period 2
Population: The rTNSS total period 2 change scores were partitioned into tertile ranges to form three groups: Low Change (-0.70 - -1.85; n = 55), Medium Change (-2.08 - -1.74; n = 56), or High Change (-6.57 - -2.14; n = 55).
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Medium Change; High Change: rTNSS change scores were partitioned into three categories to form the independent variable - Low Change (0.70 to 1.85; n = 55), Medium Change (2.08 to 1.74; n = 56), or High Change (6.57 to 2.14; n = 55) groups.
Arm/Group | Low Change | Medium Change | High Change
Number analyzed (Participants) | 54 | 56 | 55
scores on a scale
  Interference | .8838 (2.739) | 7.914 (2.195) | 6.612 (1.782)
  Regimen Adaptation | -8.462 (1.159) | -3.761 (3.447) | 4.242 (3.509)
  Role Limitation | 1.075 (1.16) | 6.079 (1.774) | 4.688 (1.465)
  Regimen Difficulty | -7.620 (2.610) | -3.751 (2.757) | .309 (2.469)
  Sensory Impact | -3.407 (3.33) | -0.500 (3.113) | 3.200 (3.172)
  Hassle | -0.648 (3.748) | 8.036 (3.052) | 10.273 (3.044)
  Burden | 1.852 (1.321) | 8.147 (2.121) | 4.602 (1.144)
  Regimen Management | 0.2521 (1.790) | 1.265 (2.156) | 1.524 (2.029)
  Perceived Relief | -6.512 (4.280) | -2.381 (3.167) | 8.424 (2.928)
  Overall Satisfaction | -2.510 (1.818) | 2.337 (1.832) | 4.875 (1.436)

5. Primary Outcome: Sensitivity Analyses of Treatment Satisfaction Subscales: Standard Effect Sizes (SES)
Description: Within-and between-responder group standardized effect sizes (SES) were calculated. The generally accepted guidelines for clinically important standard effect sizes are "small"(0.2), "medium" (0.5), and "large" (0.8).
  Between group SES indicates the magnitude of "treatment" differences. In this case, the groups were responders according to the baseline rTNSS scores. All of the treatment satisfaction subscales and satisfaction scales were scored from 0 (low satisfaction) to 100 (high satisfaction).
Time Frame: Day 1 (Pre-treatment) through Day 29
Population: Baseline rTNSS was partitioned into tertiles and patients were assigned to Low, Medium, or High symptom groups.
Measure: Number; unit: standard effect sizes
Groups:
- Low Response Group; High Response Group: Within Group Standardized Effect Sizes. TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval.
- High Minus Low Response Group: Between Group Standardized Effect Sizes. TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval.
Arm/Group | Low Response Group | High Response Group | High Minus Low Response Group
Number analyzed (Participants) | 60 | 62 | 61
standard effect sizes
  Interference | 0.551 | 0.893 | 0.474
  Regimen Adaptation | 0.057 | 0.534 | 0.553
  Role Limitation | 0.722 | 0.920 | 0.198
  Regimen Difficulty | -0.057 | 0.098 | 0.157
  Sensory Impact | 0.720 | 0.843 | 0.326
  Hassle | 0.466 | 0.926 | 0.597
  Burden | 0.898 | 0.761 | 0.064
  Regimen Management | 0.656 | 0.728 | 0.076
  Perceived Relief | -0.114 | 0.439 | 0.591

6. Primary Outcome: Principal Components Analysis (Treatment Process, Treatment Outcomes) Factor Loadings for Treatment Preference Scales
Description: Principal components analysis was conducted with varimax rotation that revealed two factors. These two factors are the principal components of the preference scale: Treatment Process and Treatment Outcomes. Loadings represent the degree each of the variables "correlates" with each of the factors. The loadings range from -1 to 1. An inspection of the factor loadings, reveals the extent to which each of the variables contributes to the meaning of each of the factors. High loading number provide meaning and interpretation of factors.
Time Frame: Day 1 (Pre-treatment) through Day 29
Population: as for outcome 1
Measure: Number; unit: factor loadings
Groups:
- Treatment Process: Extraction Method: Principal Component Analysis. Rotation Method: Varimax with Kaiser Normalization. Treatment Process Component reflects preference on items pertaining to the perceived drug treatment process, including ease of use; convenience; flexibility in daily activities; taste; use in public; smell; fewer problems with medication running out of the nose; fewer problems with medication dripping down throat; and number of sprays per dose.
- Treatment Outcomes: Extraction Method: Principal Component Analysis. Rotation Method: Varimax with Kaiser Normalization. Treatment Outcomes Component reflects the perceived outcomes of drug treatment, including longer relief; symptom relief, if both were the same price; for feeling better about your appearance; for fewer problems with irritation to nose; faster relief; and how it makes your nose feel.
Arm/Group | Treatment Process | Treatment Outcomes
Number analyzed (Participants) | 185 | 185
factor loadings
  for convenience | 0.766 | 0.433
  for ease of use | 0.764 | 0.450
  for use in public | 0.762 | 0.270
  for taste | 0.756 | 0.142
  fewer problems with medicaton running out nose | 0.722 | 0.324
  for number of sprays per dose | 0.713 | 0.331
  for flexibility in daily activities | 0.712 | 0.560
  for smell | 0.706 | 0.360
  fewer problems w/ medication dripping down throat | 0.666 | 0.234
  for longer relief | 0.230 | 0.876
  for symptom relief | 0.243 | 0.875
  for faster relief | 0.283 | 0.802
  if both were the same price | 0.433 | 0.773
  for better feeling about your appearance | 0.539 | 0.678
  for fewer problems with irritation to your nose | 0.509 | 0.587
  for how is makes your nose feel | 0.501 | 0.571

ADVERSE EVENTS:
Groups:
- Ciclesonide: ciclesonide hydrofluoroalkane nasal aerosol (HFA) 80 μg once daily pooled
- Mometasone: mometasone nasal inhalation 200 μg once daily pooled
Arm/Group | Ciclesonide | Mometasone
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/176
Other Adverse Events (participants affected / at risk) | 16/175 | 4/176
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide (N=175) | Mometasone (N=176)
Instillation Site Discomfort (General disorders) | 5 (5) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other